CLINICAL TRIAL: NCT00382395
Title: Randomized, Controlled, Multicenter Comparative Trial to Evaluate the SOLX Gold Shunt for the Reduction of Intraocular Pressure (IOP) in Glaucomatous Eyes Following Failed Medical and Conventional Surgical Treatments
Brief Title: SOLX Gold Shunt Versus Control Implant: Randomized Trial for Refractory Glaucoma
Status: Suspended | Phase: Phase 3 | Type: Interventional
Sponsor: SOLX, Inc. (Industry)
Responsible Party: Doug Adams, SOLX, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLX53
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Glaucoma; Glaucoma, Open Angle
Keywords: Glaucoma shunt; Ocular implant; Gold; trabeculectomy
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SOLX Gold Shunt
  Interventions: Device: SOLX Gold Shunt GMS-plus
- 2 (Active Comparator): Control Ahmed FP7 Shunt
  Interventions: Device: Ahmed FP7 Glaucoma Valve

INTERVENTIONS:
Device: SOLX Gold Shunt GMS-plus — Single use implant
  Arms: 1
Device: Ahmed FP7 Glaucoma Valve — Single use implant
  Arms: 2

SUMMARY:
Study Objective:

To establish the substantial equivalence of the SOLX Gold Shunt to commercially available aqueous shunts, specifically the Ahmed™ Glaucoma Valve Model FP7, in the ability to reduce intraocular pressure (IOP) associated with glaucoma in eyes where medical and conventional surgical treatments have failed.

DETAILED DESCRIPTION:
This protocol is a randomized, controlled, multi-center, outpatient study to compare the IOP lowering ability and safety profile of the SOLX Gold Shunt to the selected, commercially available aqueous shunt product (i.e., Control shunt Model FP7 Ahmed™ Glaucoma Valve Flexible Plate™) for a period of up to one year. Extended follow up is scheduled for a period not to exceed two years, should this be necessary for regulatory purposes. Follow-up beyond one year will be expected unless other patients with SOLX Gold Shunt implants in earlier phase studies outside the US clearly show no significant adverse effects associated with the long-term use of the device for follow-up periods exceeding one year, and this information is deemed adequate to reduce the required follow-up period under this protocol to a shorter period, such as 6 months for the last-to-enter patients at the time of filing for 510(k) marketing clearance review with the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Primary open-angle, pseudoexfoliative, or pigmentary glaucoma
* Age 21 or over
* refractory glaucoma, with IOP >21 mmHg on medications and failed prior incisional glaucoma surgery
* detectable visual field defect (negative MD score)
* written consent
* available for up to 24 months follow-up

Exclusion Criteria:

* either eye with VA worse than count fingers
* recent angle closure glaucoma episode
* uveitic glaucoma, iridocorneal endothelial (ICE) syndrome, traumatic glaucoma, or neovascular glaucoma
* other significant ocular disease, except cataract
* active ocular infection
* expected ocular surgery in next 12 months
* no suitable quadrant for implant
* systemic corticosteroid therapy > 5 mg/day prednisone
* intolerance to gonioscopy or other eye exams
* mental impairment interfering with consent or compliance
* pregnancy
* known sensitivity to anticipated medications used at surgery
* significant co-morbid disease
* concurrent enrollment in another drug or device study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction in IOP at both 12 and 24 months after implant | 1 & 2 years

SECONDARY OUTCOMES:
Absolute IOP | 1 & 2 years
Mean number of glaucoma medications | 1 & 2 years
Success rate | 1 & 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan S. Peterson, MS, RAC, Study Director — The Emmes Company, LLC
Locations (15):
- United States (9):
  - North Bay Eye Associates, Petaluma, California
  - Glaucoma Consultants of Colorado, Littleton, Colorado
  - International Eye Care, Tampa, Florida
  - Price Vision Group, Indianapolis, Indiana
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Glaucoma Associates of New York, New York, New York
  - Eagle Mountain Vision, Tulsa, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Tennessee / Hamilton Eye Institute, Memphis, Tennessee
- Canada (2):
  - Credit Valley EyeCare, Mississauga, Ontario
  - Institut du Glaucome de Montréal, Montreal, Quebec
- India (2):
  - Bombay City Eye Institute & Research Centre, Mumbai, Maharashtra
  - Vision Research Foundation / Sankara Nethralaya, Chennai, Tamil Nadu
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- Military Institute of the Health Services, Warsaw, Poland